CLINICAL TRIAL: NCT01614704
Title: Impact of Sequential Chemotherapy on Young Patients Breast Cancer Treated Fertility
Status: Terminated | Type: Observational
Why Stopped: End of study
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: Cancer et fertilité - 1104
Record Dates: First submitted 2012-05-18; First posted 2012-06-08 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer; Fertility
Keywords: Breast cancer; Fertility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adjuvant treatment: Patients in this group will be offered the option of ovarien cryopreservation as well as the follow up of the follicule stock during chemotherapy.
- Neo adjuvant treatment: patients in this group will only have the follow up of the follicule stock.

SUMMARY:
Breast cancer affect around 52 000 women in France each year. Amongst them, 7% are less than 40 years old and 2% are in between 25 and 35 years old. Significant therapeutic advances have improved the prognostic of these patients. They will all most likely to received chemotherapy. Despite the fact that chemotherapy has many side effects, these women do question the impact of the treatment on their ability to procreate.

On 06/08/04 law basis, each patient is allowed to preserve gametes or germinal tissues when medical care potentially affect fertility.

Functional evaluation of ovarian reserve could help comprehend new chemotherapy protocols, provide fertility information, and help individualize fertility preservation supports.

Principal objective is to ensure the absence of ovarian stimulation's side effects and assess chemotherapy effects on child carrying potential.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age < 38
* breast cancer histologically proved
* under the control of an adjuvant chemotherapy or neo adjuvant chemotherapy
* verbal agreement given

Exclusion Criteria:

* age ≥ 38
* metastatic breast cancer
* non able to follow the design of the study (geographic, social or psychological reasons)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: young female, treated for non metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
change from baseline of Anti Mullerian Hormone (AMH) rate to different time points until 24 months | baseline, Day 1 of Cycle 2, Day 1 of Cycle 4, Day 1 of Cycle 6, 3 months, 6 months, 9 months, 12 months, 24 months
  variation of percentages of AMH rate compared to baseline - Observe sequential chemotherapy on ovarian follicular content
change from baseline of account of antral follicles (CFA) rate to different time points until 24 months | baseline, Day 1 of Cycle 2, Day 1 of Cycle 4, Day 1 of Cycle 6, 3 months, 6 months, 9 months, 12 months, 24 months
  variation of percentages of CFA rate compared to baseline - Observe sequential chemotherapy on ovarian follicular content

SECONDARY OUTCOMES:
amenorrhea chemotherapeutically induced (weeks) | 4 years
  observe chemotherapy induced amenorrhea frequency and duration of amenorrhea
correlation between amenorrhea duration and oncologic outcome (overall and free disease survival) | 4 years
  collection of amenorrhea duration (weeks)
correlation between ovarian stimulation safety and oncologic outcome (overall and free disease survival) | 4 years
  toxicity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Audrey MAILLIEZ, MD, Study Chair — Oscar Lambret Center; Christine DECANTER, MD, Study Chair — CHRU LILLE
Locations (1):
- Oscar Lambret Center, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No